CLINICAL TRIAL: NCT06567769
Title: A Phase 1, Open-label, Ascending Dose Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of Recombinant Human Heparan N-Sulfatase (rhHNS, GC1130A) Via Intracerebroventricular Access Device in Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Brief Title: Phase 1 Study of GC1130A in Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC1130_MPS3A_P0101
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sanfilippo Syndrome Type A
Keywords: Mucopolysaccharidosis Type III Subtype A; MPS IIIA
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: GC1130A
- Cohort 2 (Experimental)
  Interventions: Drug: GC1130A
- Cohort 3 (Experimental)
  Interventions: Drug: GC1130A

INTERVENTIONS:
Drug: GC1130A — ICV injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of recombinant human heparan N-sulfatase (rhHNS, GC1130A) administered via intracerebroventricular access device in patients with Sanfilippo Syndrome Type A (MPS IIIA).

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented MPS IIIA diagnosis
* Participants aged ≥ 12 months and ≤ 18 years

Exclusion Criteria:

* Participants with significant non-MPS IIIA related central nervous system impairment
* Participants with previous complication from intraventricular drug administration
* Participants with contraindications for MRI scans and for neurosurgery
* Participants that received treatment with any investigational drug or a device intended as a treatment for MPS IIIA within 30 days or 5 half-lives prior to the study
* Participants that received a hematopoietic stem cell or bone marrow transplant or received gene therapy

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidences and characteristics of adverse events | up to 108 weeks

SECONDARY OUTCOMES:
Maximum concentration in cerebrospinal fluid (CSF) | up to 104 weeks
  GC1130A PK parameters
Area under the concentration-time curve in CSF | up to 104 weeks
  GC1130A PK parameters
Maximum concentration in serum | up to 104 weeks
  GC1130A PK parameters
Area under the concentration-time curve in serum | up to 104 weeks
  GC1130A PK parameters
Change from baseline in CSF heparan sulfate concentration | up to 104 weeks
Change from baseline in serum heparan sulfate concentration | up to 104 weeks
Incidence of anti-drug and neutralizing antibodies of GC1130A in CSF | up to 104 weeks
Incidence of anti-drug and neutralizing antibodies of GC1130A in serum | up to 104 weeks
Change from baseline in raw scores in cognitive domain of Bayley Scales of Infant and Toddler Development Scores-3rd edition (BSID-III) | up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - UCSF Benioff Children's Hospital, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota
- National Center for Child Health and Development, Setagaya City, Tokyo, Japan
- South Korea (2):
  - Ajou University Medical Center, Suwon, Gyeongi-do
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No